CLINICAL TRIAL: NCT06998641
Title: EFFECTİVİTY OF CHITOSAN COVERED GAUZE IN POSTPARTUM HEMORRHAGIC OBSTETRIC LACERATIONS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Doruk Cevdi Katlan, Maternal Fetal Medicine Specialist, Istanbul Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISTANBUL TRH - 21.03.2025 - 65
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Effectiveness of Chitosan Covered Gauze to Stop Bleeding in Post-partum Tears; Comparison of the Effect of Chitosan Covered Gauze With Suturing in Terms of Hemostasis in Post-partum Haemorrhagic Tears
Keywords: chitosan-covered-gauze; post-partum lacerations; obstetrical tears

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chitosan-covered-gauze applied tears (Experimental): Hemostasis of the tears is obtained by the application of chitosan-covered-gauze
  Interventions: Procedure: Chitosan-covered-gauze application
- Suturation group (Active Comparator): Hemostasis of the tears is obtained by suturing
  Interventions: Procedure: Suturation

INTERVENTIONS:
Procedure: Chitosan-covered-gauze application — Effectiveness of chitosan-covered-gauze in terms of patients' comfort and satisfaction, hospital stay, total amount of bleeding, hemoglobin decline and other complications (infections, need for transfusion etc.) for the treatment of hemorrhagic obstetrical tears
  Arms: chitosan-covered-gauze applied tears
Procedure: Suturation — Effectiveness of suturation in terms of patients' comfort and satisfaction, hospital stay, total amount of bleeding, hemoglobin decline and other complications (infections, need for transfusion etc.) for the treatment of hemorrhagic obstetrical tears
  Arms: Suturation group

SUMMARY:
This study was planned to investigate the efficacy of different treatment methods that can be used in the treatment of hemorrhagic tears that may occur in the postpartum period. The volunteers who will participate in the study will be evaluated during the hospitalization period after delivery and at the end of the puerperium 6 weeks after delivery, in accordance with routine postpartum control examinations. In the treatment of postpartum hemorrhagic tears, the treatment options such as suturing the tears to stop bleeding or applying tampons with bleeding stopping agent (chitosan) and compression effect to the torn area will be determined completely randomly.

ELIGIBILITY:
Inclusion Criteria: Patients, 18-48 years old, who gave birth in Istanbul TRH between March 2025 and March 2027 experiencing 1st and 2nd degree obstetric lacerations with postpartum hemorrhage without the need for anatomical defect repairing and without additional conditions such as uterine atony, placental rest, etc. that may affect the amount of postpartum bleeding.

Exclusion Criteria: Patients not fullfilling the inclusion criteria in terms of age limits, time and place of birth or ones who are experiencing 1st and 2nd degree obstetric lacerations with postpartum hemorrhage with the need for anatomical defect repairing and with additional conditions such as uterine atony, placental rest, etc. that may affect the amount of postpartum bleeding.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 62 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Amount of bleeding | From time of birth to the cessation of bleeding
  Total amount of blood which is calculated by subtracting the dry weight of surgical absorbant gauze materials from their soaked weight

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Training and Research Hospital Department of Obstetrics and Gynecology, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided